CLINICAL TRIAL: NCT01838746
Title: Percutaneous Coronary Intervention Versus Coronary Artery Bypass Grafting in Patients Aged < 50 Years: a Multicenter Study
Brief Title: CRAGS (Coronary aRtery diseAse in younG adultS)
Acronym: CRAGS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Collaborators: Finnish Foundation for Cardiovascular Research (Other)
Responsible Party: Principal Investigator, Fausto Biancari, MD, MD, PhD, University of Turku
Other Study IDs: CRAGS-1
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndromes; Young Patient; Percutaneous Coronary Intervention; Coronary Artery Bypass Grafting
Keywords: Percutaneous coronary intervention; Coronary artery bypass grafting; Coronary artery bypass surgery; Survival; Acute coronary syndrome; ST segment elevation myocardial infarction; Non-ST segment elevation myocardial infarction; Younge patient
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCI: Patients undergoing PCI
- CABG: Patients undergoing CABG

SUMMARY:
Young patients requiring myocardial revascularization are generally considered at low operative risk, but data on their immediate and late outcome are scarce. The decision-making process in these young patients is complicated by the potentially aggressive nature of premature coronary artery disease and their likely long expectancy of life, which expose them to a significantly higher risk of recurrent coronary events as well as the need of repeat revascularization. The lack of data on long-term outcome as well as on operative details (in particular, on the use of arterial grafts) and peri- and postoperative medication prevent any conclusive results on the durability either of coronary artery bypass grafting (CABG) or of percutaneous coronary intervention (PCI) in these young patients. Furthermore, recent advances in stents technology as well in peri- and postoperative medical treatment indicate the need a comparative study to define the baseline characteristics of patients aged < 50 years undergoing either PCI or CABG and to evaluate their current immediate and late outcome.

DETAILED DESCRIPTION:
Age is, without any doubt, one of the most important risk factors for adverse events after any cardiovascular procedure and because of this it is incorporated in all major risk scoring methods. There is abundant literature dealing with the outcome of elderly patients undergoing cardiovascular procedures as their operative risk is significantly increased and preoperative risk assessment is of great importance in the decision-making process of these fragile patients (1). In the very elderly patients percutaneous coronary intervention (PCI) is an attractive treatment method, particularly in those with multiple comorbidities (2). On the other hand, coronary artery bypass grafting (CABG) has been shown to be a durable procedure also among octogenarians (2).

Young patients requiring myocardial revascularization are generally considered at low operative risk, but data on their immediate and late outcome are scarce. However, the decision-making process in these young patients is complicated by the potentially aggressive nature of premature coronary artery disease and their likely long expectancy of life, which expose them to a significantly higher risk of recurrent coronary events as well as the need of repeat revascularization. CABG seems to more durable compared with percutaneous coronary intervention (3), particularly because of excellent late results with the use arterial grafts (4). Therefore, young patients with diffuse coronary artery diffuse may likely benefit of surgical revascularization. However, no formal comparative analysis of these two treatment methods has been previously performed in this young patient population. Since CABG is a major procedure with a potential risk of operative mortality and major morbidity, this is an argument against surgical revascularization, even if recent pooled data showed that it can be performed with an exceedingly low mortality risk (0.9%) (Biancari et al. submitted, Fig. 1).

Such a low postoperative mortality rate is similar to that reported by Khawaja et al. (5) in patients aged ≤ 50 years treated by PCI (0.86%). However, PCI was performed in 41% of these patients with single vessel coronary artery disease. This is likely to significantly differ from surgical series (6).

Only two studies evaluated the outcome after CABG in patients aged < 40 years (7) and < 50 years (8) and estimated a survival rate at 10 years of about 75%. A study by Ellis (9) addressed survival after PCI in 86 patients aged < 40 years and showed a 10-year survival rate of about 91%, but a significant number of patients underwent repeat PCI (37%) and/or CABG (22%). These findings should be viewed in the light of the fact that most of patients did not have diffuse coronary artery disease (3-vessel disease was present in 11% of patients) and they were treated about two decades ago. Khawaja et al. (6) reported on 2922 patients aged ≤ 50 years who underwent percutaneous coronary intervention since 1979 and having a 5-year survival of about 95%. They reported repeat target revascularization rates ranging from 19% to 27% according to different study periods.

The lack of data on long-term outcome as well as on operative details (in particular, on the use of arterial grafts) and peri- and postoperative medication prevent any conclusive results on the durability either of CABG of PCI in these young patients. Furthermore, recent advances in stents technology as well in peri- and postoperative medical treatment indicate the need a comparative study to define the baseline characteristics of patients aged < 50 years undergoing either PCI or CABG and to evaluate their current immediate and late outcome.

ELIGIBILITY:
Inclusion Criteria:

- age < 50

Exclusion Criteria:

* age > 50

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged < 50 years who underwent CABG or PCI from 2005 to 2012 will be collected from multiple institutions.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Repeat revascularization | Three years
  Any percutaneous coronary intervention or coronary artery bypass grafting after primary revascularization

SECONDARY OUTCOMES:
All-cause mortality | Three years
Major cardiovascular and cerebral events (MACCE) | Three years
Stroke | Three years
Myocardial infarction | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Biancari, MD, PhD, Principal Investigator — Oulu University Hospital; Juhani Airaksinen, MD, PhD, Study Chair — Turku University Hospital
Locations (9):
- Finland (5):
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa
- University of Iceland, Reykjavik, Iceland
- Italy (2):
  - University of Catania, Catania
  - University of Verona Medical School, Verona
- Sahlgrenska Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Gunn J, Kuttila K, Vasques F, Virtanen R, Lahti A, Airaksinen J, Biancari F. Comparison of results of coronary artery bypass grafting versus percutaneous coronary intervention in octogenarians. Am J Cardiol. 2012 Oct 15;110(8):1125-9. doi: 10.1016/j.amjcard.2012.05.055. Epub 2012 Jul 3. PMID 22762714
- [Background] Nissinen J, Wistbacka JO, Loponen P, Korpilahti K, Teittinen K, Virkkila M, Tarkka M, Biancari F. Coronary artery bypass surgery in octogenarians: long-term outcome can be better than expected. Ann Thorac Surg. 2010 Apr;89(4):1119-24. doi: 10.1016/j.athoracsur.2009.12.063. PMID 20338317
- [Background] Kappetein AP, Feldman TE, Mack MJ, Morice MC, Holmes DR, Stahle E, Dawkins KD, Mohr FW, Serruys PW, Colombo A. Comparison of coronary bypass surgery with drug-eluting stenting for the treatment of left main and/or three-vessel disease: 3-year follow-up of the SYNTAX trial. Eur Heart J. 2011 Sep;32(17):2125-34. doi: 10.1093/eurheartj/ehr213. Epub 2011 Jun 22. PMID 21697170
- [Background] Locker C, Schaff HV, Dearani JA, Joyce LD, Park SJ, Burkhart HM, Suri RM, Greason KL, Stulak JM, Li Z, Daly RC. Multiple arterial grafts improve late survival of patients undergoing coronary artery bypass graft surgery: analysis of 8622 patients with multivessel disease. Circulation. 2012 Aug 28;126(9):1023-30. doi: 10.1161/CIRCULATIONAHA.111.084624. Epub 2012 Jul 18. PMID 22811577
- [Background] Cole JH, Miller JI 3rd, Sperling LS, Weintraub WS. Long-term follow-up of coronary artery disease presenting in young adults. J Am Coll Cardiol. 2003 Feb 19;41(4):521-8. doi: 10.1016/s0735-1097(02)02862-0. PMID 12598059
- [Background] Canver CC, Nichols RD, Cooler SD, Heisey DM, Murray EL, Kroncke GM. Influence of increasing age on long-term survival after coronary artery bypass grafting. Ann Thorac Surg. 1996 Oct;62(4):1123-7. doi: 10.1016/0003-4975(96)00446-8. PMID 8823100
- [Background] Ellis CJ, French JK, White HD, Ormiston JA, Whitlock RM, Webster MW. Results of percutaneous coronary angioplasty in patients <40 years of age. Am J Cardiol. 1998 Jul 15;82(2):135-9. doi: 10.1016/s0002-9149(98)00318-x. PMID 9678280
- [Derived] Lautamaki A, Airaksinen KE, Kiviniemi T, Vinco G, Ribichini F, Gunn J, Anttila V, Heikkinen J, Korpilahti K, Karjalainen P, Kajander O, Eskola M, Ilveskoski E, Axelsson T, Gudbjartsson T, Jeppsson A, Biancari F. Prognosis and disease progression in patients under 50 years old undergoing PCI: the CRAGS (Coronary aRtery diseAse in younG adultS) study. Atherosclerosis. 2014 Aug;235(2):483-7. doi: 10.1016/j.atherosclerosis.2014.05.953. Epub 2014 Jun 9. PMID 24953487
- [Derived] Biancari F, Gudbjartsson T, Heikkinen J, Anttila V, Makikallio T, Jeppsson A, Thimour-Bergstrom L, Mignosa C, Rubino AS, Kuttila K, Gunn J, Wistbacka JO, Teittinen K, Korpilahti K, Onorati F, Faggian G, Vinco G, Vassanelli C, Ribichini F, Juvonen T, Axelsson TA, Sigurdsson AF, Karjalainen PP, Mennander A, Kajander O, Eskola M, Ilveskoski E, D'Oria V, De Feo M, Kiviniemi T, Airaksinen KE. Comparison of 30-day and 5-year outcomes of percutaneous coronary intervention versus coronary artery bypass grafting in patients aged</=50 years (the Coronary aRtery diseAse in younG adultS Study). Am J Cardiol. 2014 Jul 15;114(2):198-205. doi: 10.1016/j.amjcard.2014.04.025. Epub 2014 May 2. PMID 24878127